CLINICAL TRIAL: NCT07283419
Title: Family Environment and Cognitive Function as Predictors of Efficacy for rTMS Combined With Group Therapy in Adolescent Depression: A Prospective Cohort Study
Brief Title: Predictors of rTMS and Group Therapy Efficacy in Adolescent Depression
Status: Completed | Type: Observational
Sponsor: The First Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Yanju Liu, Principal investigator, The First Hospital of Hebei Medical University
Other Study IDs: 2023S00133
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Major Depressive Disorder (MDD); Adolescent Depression
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- rTMS + Group Therapy Cohort: Adolescents diagnosed with MDD who received the standardized combined intervention.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS); Behavioral: Group Cognitive Behavioral Therapy (CBT)

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — High-frequency (10 Hz) rTMS applied over the left dorsolateral prefrontal cortex (DLPFC), administered 5 days per week for 4 weeks (20 sessions total).
Behavioral: Group Cognitive Behavioral Therapy (CBT) — Manualized group therapy sessions focused on psychoeducation, cognitive restructuring, emotion regulation, and interpersonal skills, held twice weekly for 4 weeks (8 sessions total).

SUMMARY:
This study aims to identify baseline predictors of treatment efficacy in adolescents with Major Depressive Disorder (MDD) undergoing a combined intervention of repetitive transcranial magnetic stimulation (rTMS) and group therapy. Specifically, the study investigates the predictive value of family environment characteristics (cohesion, conflict, expressiveness) and cognitive functions (executive function, attention/inhibition).

DETAILED DESCRIPTION:
Adolescent depression is a significant health concern, and while combined therapies involving neuromodulation and psychotherapy show promise, individual treatment responses vary heterogeneity. This prospective cohort study enrolled 163 adolescents aged 12-18 with MDD. All participants received a standardized 4-week intervention consisting of 20 sessions of high-frequency (10 Hz) rTMS over the left dorsolateral prefrontal cortex (DLPFC) and 8 sessions of group Cognitive Behavioral Therapy (CBT).

Baseline assessments included the Family Environment Scale (FES) and a neuropsychological battery including the Stroop Color-Word Test and Wisconsin Card Sorting Test (WCST). The primary outcome was the percentage reduction in depressive symptoms measured by the HAMD-24 scale. The study employs multiple linear regression to determine which baseline factors independently predict superior treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of Major Depressive Disorder (MDD) according to ICD-10 criteria.
* Score of ≥ 20 on the 24-item Hamilton Depression Rating Scale (HAMD-24).
* Sufficient intellectual and linguistic ability to complete assessments and participate in therapy.
* Provided written informed consent (participants and guardians).

Exclusion Criteria:

* Lifetime diagnosis of a psychotic or bipolar disorder.
* Current substance use disorder.
* Significant neurological illness (e.g., epilepsy) or metallic implants contraindicated for rTMS.
* Receiving concurrent formal psychotherapy outside the study protocol.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Inpatients aged 12 to 18 years recruited from the Department of Mental Health at The First Hospital of Hebei Medical University between August 2023 and July 2024. All participants had a primary diagnosis of Major Depressive Disorder (MDD) according to ICD-10 criteria and received a standardized combined intervention of rTMS and group therapy.
Sampling Method: Non-Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Percentage Reduction in HAMD-24 Score | Baseline and Week 4
  Treatment efficacy is defined as the percentage reduction in the 24-item Hamilton Depression Rating Scale (HAMD-24) score from baseline to the end of treatment. The formula used is: [(HAMD-24 at Baseline - HAMD-24 at Week 4) / HAMD-24 at Baseline] × 100%. The HAMD-24 assesses the severity of depressive symptoms, with higher scores indicating more severe depression.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Hebei Medical University, Shijiazhuang, Hebei, China